CLINICAL TRIAL: NCT03422978
Title: Anesthetic Sparing Effect of Dexmedetomidine During TIVA With Propofol and Remifentanil for Children Undergoing Dental Procedures
Brief Title: The Effects of Dexmedetomidine on Intravenous Anesthetic Requirements for Children Undergoing Dental Procedures
Acronym: Dexmed-PRS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Simon Whyte, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: H17-02157
Record Dates: First submitted 2017-12-08; First posted 2018-02-06 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Anesthetic Sparing
Keywords: Dexmedetomidine
MeSH Terms: interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessor of sedation scores post-procedure will be blinded to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Saline bolus (Sham Comparator): 10mL normal saline solution administered intravenously over 60 seconds starting after intubation.
  Interventions: Drug: Normal saline
- Dexmedetomidine 0.25 mcg/kg (Experimental): 0.25 mcg/kg dexmedetomidine diluted with normal saline to a 10mL volume, administered intravenously over 60 seconds starting after intubation.
  Interventions: Drug: Dexmedetomidine
- Dexmedetomidine 0.50 mcg/kg (Experimental): 0.50 mcg/kg dexmedetomidine diluted with normal saline to a 10mL volume, administered intravenously over 60 seconds starting after intubation.
  Interventions: Drug: Dexmedetomidine
- Dexmedetomidine 1.00 mcg/kg (Experimental): 1.00 mcg/kg dexmedetomidine diluted with normal saline to a 10mL volume, administered intravenously over 60 seconds starting after intubation.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Single dose dexmedetomidine administered over 60 seconds post-induction.
  Other Names: Precedex
  Arms: Dexmedetomidine 0.25 mcg/kg; Dexmedetomidine 0.50 mcg/kg; Dexmedetomidine 1.00 mcg/kg
Drug: Normal saline — Single dose normal saline administered over 60 seconds post-induction.
  Arms: Saline bolus

SUMMARY:
The investigators propose to determine the propofol and remifentanil sparing effects of a single dose of dexmedetomidine in the dental population. The investigators plan to do this by performing a blinded study with 4 test groups (3 experimental and 1 control), using BIS monitoring to titrate TIVA infusion to an acceptable depth of anesthesia.

DETAILED DESCRIPTION:
Purpose:

To determine an optimal dose of dexmedetomidine for its anesthetic sparing effect, without extending post-operative stay.

Hypothesis:

The investigators hypothesize that dexmedetomidine will cause a clinically significant reduction of 30% in the amount of propofol and remifentanil required to maintain adequate depth of anesthesia, as monitored through the Bispectral Index.

Justification:

The dose-sparing effect of dexmedetomidine on TIVA requirements and the dose-response relationship between dexmedetomidine and TIVA dosing regimens has not been explored in young children. This study will have many relevant applications to many areas of pediatric anesthesia practice, such as craniofacial and neurosurgery, sedation techniques in diagnostic and interventional radiology, out of OR sedation, and in all young children in whom minimizing anesthesia exposure is increasingly sought given possible concerns over the long term neurocognitive effects of surgery and anesthesia in early life.

Objectives:

To investigate the dose-sparing effect on a propofol/remifentanil infusion of bolus doses of dexmedetomidine and to characterize the dose-response relationship between dexmedetomidine doses and TIVA dose reduction.

Research Design:

The investigators propose a randomized, 4-group comparative study to characterize the effects of different bolus doses of dexmedetomidine on the infusion requirements of propofol and remifentanil. The study-specific interventions will include a bolus of dexmedetomidine (or placebo) at induction of anesthesia, and maintenance of anesthesia, titrated to a Bispectral index of 50-60, with propofol and remifentanil infusions.

Statistical Analysis:

Standard statistical analysis will be undertaken using R Foundation for Statistical Computing, Vienna, Austria). Summary data will be tabulated and presented as median (IQR). Mean infusion rates of propofol and remifentanil will be compared between groups using Wilcoxon signed-rank test, with 95% confidence intervals obtained by the Hodges-Lehmann estimator. Dose (in mcg/kg) of additional opioids given in PACU will be tabulated and compared using Fisher's exact test. Bonferroni corrections will be applied as appropriate whenever multiple comparisons are performed.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2
* Elective dental surgery
* Planned general anesthesia with TIVA
* Age 2-10 years

Exclusion Criteria:

* General anesthesia with inhalation induction
* Documented seizure disorder
* Cardiac disease
* Cardiac rhythm abnormalities
* Chronic hypertension
* Weight < 5th centile or > 95th centile for age
* Pre-operative administration of anxiolytics (such as benzodiazepines or opioid analgesics)
* Hypersensitivity to dexmedetomidine or any other study medication

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Propofol and remifentanil sparing | Through length of procedure, an average of 1.5 hours
  Propofol and remifentanil sparing as measured by time-averaged, total administered doses of propofol (mg/kg) and remifentanil (mcg/kg) compared to the placebo group.
Propofol and remifentanil infusion rate reduction | Through length of procedure, an average of 1.5 hours
  Change in infusion rates of propofol and remifentanil (in micrograms/kg/min), measured over time compared to the placebo group.

SECONDARY OUTCOMES:
PACU sedation | 30min post-procedure
  Sedation will be scored from 0 (alert) to 4 (unarousable) using the University of Michigan sedation score (UMSS) at 10, 20, and 30 minutes post discontinuation of the infusions.
PACU pain scores | 30min post-procedure
  Pain will be scored from 0 (no pain) to 10 (severe pain), using the FLACC pain scale for ages 2-7 and the FACES pain scale for ages 8-10, and total fentanyl doses in mcg/kg given in the Post Anesthetic Care Unit will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Whyte, MBBS, FRCA, Principal Investigator — BC Children's Hospital, Department of Anesthesia
Locations (1):
- BC Children's Hospital - Department of Anesthesia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee VCL, Ridgway R, West NC, Gorges M, Whyte SD. Anesthetic-sparing effect of dexmedetomidine during total intravenous anesthesia for children undergoing dental surgery: A randomized controlled trial. Paediatr Anaesth. 2024 Dec;34(12):1213-1222. doi: 10.1111/pan.14987. Epub 2024 Aug 28. PMID 39193655
- See also: Pediatric Anesthesia Research Team website — http://part.bcchr.ca/